CLINICAL TRIAL: NCT03613532
Title: A Phase 1 Study of Adding Venetoclax to a Reduced Intensity Conditioning Regimen and to Maintenance in Combination With a Hypomethylating Agent After Allogeneic Hematopoietic Cell Transplantation for Patients With High Risk AML, MDS, and MDS/MPN Overlap Syndromes
Brief Title: Venetoclax Added to Fludarabine + Busulfan Prior to Transplant and to Maintenance Therapy for AML, MDS, and MDS/MPN
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jacqueline Garcia, MD (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Jacqueline Garcia, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-283
Record Dates: First submitted 2018-07-26; First posted 2018-08-03 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS); Chronic Myelomonocytic Leukemia (CMML); MDS/Myeloproliferative Neoplasm-unclassifiable (MDS/MPN-unclassifiable); Hematopoietic Stem Cell Transplant
Keywords: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS); Chronic Myelomonocytic Leukemia (CMML); MDS/myeloproliferative neoplasm-unclassifiable (MDS/MPN-unclassifiable); Hematopoietic Stem Cell Transplant
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — venetoclax; fludarabine; fludarabine phosphate; Busulfan; Azacitidine; decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Venetoclax (Experimental): Part 1 dose escalation
  * Venetoclax: 6-7 total doses based on level assigned
  * Busulfan: given 2x daily for 4 days
  * Fludarabine: given 1x daily for 4 days Part 2 includes post-transplant therapy with azacitidine and venetoclax for 8-12 cycles per dose level.
  Part 3 includes post-transplant therapy with oral decitabine/cedazuridine and venetoclax for 8 cycles.
  Part 4 assesses PTCy/Tac/MMF GVHD regimen instead of Tac/Methotrexate -post transplant period includes therapy with azacitidine and venetoclax for 8 cycles.
  Interventions: Drug: Venetoclax; Drug: Fludarabine; Drug: Busulfan; Drug: Azacitidine; Drug: Decitabine/cedazuridine

INTERVENTIONS:
Drug: Venetoclax — Part 1: 6-7 total doses depending on dose level assigned
  Other Names: ABT199
Drug: Fludarabine — Given once daily for 4 days
  Other Names: Fludara
Drug: Busulfan — Given twice daily for 4 days
  Other Names: Busulfex; Myleran
Drug: Venetoclax — Part 2, Part 3, and Part 4: 14 doses for 8-12 cycles depending on dose level assigned
  Other Names: ABT199
Drug: Azacitidine — Part 2 and Part 4: 5 doses for 8-12 cycles depending on dose level assigned
Drug: Decitabine/cedazuridine — Part 3: 3 doses for 8 cycles

SUMMARY:
This clinical trial involves individuals who have been diagnosed with Acute Myeloid Leukemia (AML), Myelodysplastic Syndrome (MDS), Chronic Myelomonocytic Leukemia (CMML), or MDS/myeloproliferative neoplasm-unclassifiable (MDS/MPN-unclassifiable) and are planning to have an allogeneic hematopoietic stem cell transplant ("bone marrow transplant"). The goal of this research study is to (1) test the safety of adding the study drug, Venetoclax, to a standard of care conditioning regimen for bone marrow transplantation as a possible means of eliminating residual (left-over) disease prior to transplant, (2) to test the safety of combination Venetoclax and azacitidine as "maintenance therapy" after transplant to possibly prevent disease recurrence and (3) to test the safety of combination Venetoclax and oral decitabine/cedazuridine as "maintenance therapy" after transplant to possibly prevent disease recurrence.

* The name of the study drug involved in this study is Venetoclax.
* It is expected that about 102 people will take part in this research study.

DETAILED DESCRIPTION:
* This research study is a Phase I clinical trial, which tests the safety of an investigational drug and tries to define the appropriate dose and schedule of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.
* There are four parts to this research study:

  * Part 1 is to determine a safe dose of the study drug, Venetoclax, when given in combination with a standard chemotherapy. Part 2 is to determine the safety of post-transplant maintenance therapy with the combination of azacitidine and venetoclax. Part 3 is to determine the safety of post-transplant maintenance therapy with the combination of oral decitabine/cedazuridine and venetoclax. Part 4 is to determine the safety of adding venetoclax to FluBu2/ post-transplant cyclophosphamide/ tacrolimus/ mycophenolate mofetil for patients undergoing RIC allo-HCT.
  * Participants enrolled in Part 1 of this study, will receive Venetoclax in combination with conditioning chemotherapy (prior to transplantation).
  * Participants enrolled in Part 2, Part 3, and Part 4 of the study, will also receive Venetoclax in combination with conditioning chemotherapy (prior to transplantation) and will have the opportunity to receive maintenance chemotherapy (after transplantation) for potentially a year.
* Part 1, Part 2, and Part 3 of this research study will have a Dose-Escalation phase. The Dose-Escalation phase is the part of the study where treatment dose and schedule are being tested.

  * In Part 1, the Dose-Escalation phase is when venetoclax will be given at different doses until the safest maximum dose has been identified. Part 1 also includes a second phase of the study which is called the Dose-Expansion phase, during which more participants will be treated at this dose level to obtain additional information on safety.
  * In Part 2, the Dose-Escalation phase is where the combination of venetoclax and azacitidine will be given after transplantation at different schedules.
  * In Part 3, the Dose-Escalation phase is where the combination of venetoclax and oral decitabine/cedazuridine will be given after transplantation at different schedules.
  * For both the Dose-Escalation or Dose-Expansion phase of this study, there will be a screening period, a pre-transplant period, a transplant period, and a post-transplant follow up period.
* In this research study, participants will receive venetoclax plus chemotherapy. Participants in Part 1, Part 2, Part 3, and Part 4 of this study will receive chemotherapy immediately prior to transplantation, which is called the "conditioning regimen." The conditioning regimen chemotherapy will suppress the immune system and may help to destroy cancer cells. During this process normal bone marrow cells are destroyed as well, thus making way for donor stem cells.

  * Fludarabine and busulfan (FluBu2) are both chemotherapies and a common conditioning regimen.
  * In this study, Venetoclax is added to the conditioning regimen (FluBu2) prior to transplantation to eliminate leftover blood cancer cells prior to transplant.
  * Participants in Part 2 and Part 4 of the study will also have the opportunity to receive venetoclax plus azacitidine after transplantation. The combination of these two drugs is called "maintenance therapy," which is treatment given after transplant to potentially reduce the chance of disease relapse. Relapse is a cause of transplant failure and can occur when there are leftover blood cancer cells.
  * Participants in Part 3 of the study will also have the opportunity to receive venetoclax plus oral decitabine/cedazuridine after transplantation. The combination of these two drugs is called "maintenance therapy," which is treatment given after transplant to potentially reduce the chance of disease relapse. Relapse is a cause of transplant failure and can occur when there are leftover blood cancer cells.
* The FDA (U.S. Food and Drug Administration) has approved Venetoclax in combination with cytarabine, azacitidine or decitabine for the treatment of newly diagnosed acute myeloid leukemia, but not for use in with conditioning chemotherapy prior to transplantation or after transplant with maintenance chemotherapy. Venetoclax is an oral drug that selectively inhibits Bcl-2, which is critical for keeping cancer cells alive.

ELIGIBILITY:
Part 1 Inclusion Criteria:

* Age 18 years and older.
* Patients must have a prior diagnosis of one of the following:

  * (Note: Mutational and cytogenetic studies performed at sites other than Dana-Farber Cancer Institute or Brigham and Women's Hospital will require review of the outside cytogenetic and/or molecular pathology reports by the overall PI.)

    * High-risk MDS, which is defined as one of the following subsets:

      * IPSS Intermediate-2 or higher
      * Presence of a mutation in TP53
      * Prescence of mutation in the RAS pathway including NRAS, KRAS, PTPN11, CBL, NF1, RIT1, FLT3, and KIT
      * Therapy-related MDS
    * High-risk AML, which is defined as one of the following subsets:

      * AML with adverse risk disease according to ELN guidelines including one of the following features:

        * a history of mutation in TP53, RUNX1, or ASXL1
        * t(6;9)(p23;q34.1); DEK-NUP214
        * t(v;11q23.3); KMT2A rearranged
        * t(9;22)(q34.1;q11.2); BCR-ABL1
        * inv(3)(q21.3q26.2) or t(3;3)(q21.3;26.2); GATA2,MECOM(EVI1)
        * -5 or del(5q)
        * -7
        * -17/abn(17p)
        * Complex karyotype
        * Monosomal karyotype
        * Wild-type NPM1 and FLT3-ITDhigh
      * Secondary AML, which is defined as a history of antecedent hematologic disorder (an MPN or MDS), a diagnosis of therapy-related myeloid neoplasm including t-MDS and t-AML, or AML with myelodysplasia-related changes, OR
      * "Secondary-type" AML, which is defined by the presence of a mutation in any of the following eight genes with high specificity for the presence of antecedent myelodysplastic syndrome including SRSF2, SF3B1, U2AF1, ZRSR2, ASXL1, EZH2, BCOR, or STAG2
      * Patients with AML with evidence of measurable residual disease by multiparameter flow cytometry (≥ 0.1%) despite morphologic remission on the pre-transplant/screening bone marrow biopsy. Review required by overall PI.
    * High-risk chronic myelomonocytic leukemia (CMML) or MDS/MPN unclassifiable (MDS/MPN-U), which is defined by the presence of trisomy 8, chromosome 7 abnormalities or complex karyotype (3 or more abnormalities); or by the presence of a mutation in ASXL1
  * Measurable disease is not required for eligibility.
  * Patient is determined to be a suitable candidate for an allo-HCT using a reduced intensity conditioning (RIC) regimen using peripheral blood stem cell as stem cell source.
  * Patient must have a matched related or an 8/8 unrelated donor option for his/her allo-HCT.
  * Patient must have an ECOG performance status ≤ 2
  * There are no limitations or minimum on the amount of prior therapy for patient's advanced myeloid malignancy. Prior exposure to venetoclax is allowed.
  * Patient must have normal organ function as defined below:

    * Total bilirubin ≤ 2.0 x institutional upper limit of normal (In patients with Gilbert's Syndrome, Total Bilirubin ≥ 2.0 is permitted.)
    * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional upper limit of normal
    * Creatinine clearance ≥ 30 mL/min using Cockcroft Gault formula
  * The effects of venetoclax on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of venetoclax administration. For women who are of child-bearing potential, they must have a negative serum beta-HCG (human chorionic gonadotropin) test to be eligible.
  * Ability to understand and the willingness to sign a written informed consent document

Part 1 Exclusion Criteria:

* Patients who have had chemotherapy (with the exception of hydroxyurea and/or dexamethasone) or radiotherapy or investigational therapy within 14 days prior to starting treatment on study. Exceptions: Patients already on venetoclax therapy prior to transplant need a three day wash out prior to first treatment dose on study. Patients on BCR-ABL, IDH and FLT3 small molecule inhibitors can stay on this treatment up until 5 days prior to first treatment dose on study.
* Patients with > 10% morphologic blasts on bone marrow biopsy if they have a diagnosis of MDS or MDS/MPN. Patients > 5% morphologic blasts on bone marrow biopsy if they have a diagnosis of AML.
* Patients recommended to receive a myeloablative conditioning regimen prior to transplantation (since there is a known survival advantage for AML using higher intensity).
* Patients who have a history of prior allogeneic stem cell transplantation.
* Symptomatic or untreated known CNS involvement of disease
* Patients with active heart disease (New York Heart Association class 3-4 as assessed by history and physical exam, or a critical event including unstable angina/stroke/myocardial infarction within the last 6 months prior to first dose on study).
* Patients who have consumed grapefruit, grapefruit products, Seville oranges or starfruit within 3 days prior to study treatment. Patients who a strong or moderate inducer within 7 days prior to the first dose of study drug.
* Malabsorption syndrome or other clinically significant condition that would preclude enteral administration.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the patient inappropriate for enrollment into this study.
* Patients with known active hepatitis B virus (HBV) infection should be excluded because of potential effects on immune function and/or drug interactions. However, if a patient has HBV history with an undetectable HBV load by polymerase chain reaction (PCR), no liver-related complications, and is on definitive HBV therapy that is not contraindicated on this study, then he/she would be eligible for study.
* Patients with known active hepatitis C virus (HCV) infection. However, if a patient with a history of HCV infection has received definitive therapy (and is now HCV viral load negative), or if a patient has a reactive HCV antibody test but has an undetectable viral load by PCR, then he/she would be eligible.
* Patients with known active HIV infection out of concern for the drug-drug interaction with venetoclax and HAART therapy.
* Pregnant or breastfeeding women or those intending to become pregnant during the study or within 3 months after the final dose of study treatment are excluded from this study. Women of childbearing potential must have a negative serum pregnancy test resulted during screening and repeated within 7 days prior to study drug (local labs are allowed).
* Vaccination with live, attenuated vaccines within 4 weeks prior to initiation of study treatment or anticipation of need for such a vaccine during the study.
* Patients with uncontrolled infection at time of first dose of treatment on study. Patients receiving anti-microbial agents including antibiotics, antiviral and antifungal therapies are allowed if hemodynamically stable.
* Part 2, Part 3, and Part 4 only: Patients recommended to receive FLT3 inhibitor therapy or any other antileukemic therapy for AML as maintenance post allo-HCT.

Part 2 and Part 3 Eligibility Criteria:

* No DLT event (including delay in neutrophil engraftment) due to the addition of venetoclax to conditioning chemotherapy prior to start of maintenance therapy.
* No morphologic evidence of relapse (defined as 5% or more morphologic blasts) prior to start of maintenance therapy confirmed by bone marrow biopsy after day +28.
* ANC ≥ 1.0 K/uL without growth factor support and platelet level ≥ 50 K/uL without platelet transfusion within 7 days of starting maintenance therapy.

  --Exception: Patients without morphologic evidence of disease relapse but with evidence of persistent molecular or cytogenetic residual disease at the time of assessment can start maintenance therapy as long as ANC ≥ 0.75 K/uL without growth factor support and platelet level ≥ 25 K/uL.
* Absence of overall grade II-IV acute GVHD per investigator. Upon acute GVHD resolution, patients are eligible. Patients that are on prednisone 0.5 mg/kg daily dose or lower are allowed to initiate maintenance.
* Total bilirubin less than or equal to 2 x institutional ULN (unless has known Gilbert's disease).
* AST and ALT less than or equal to 3 x ULN.
* Cr Cl ≥ 30 mL/min or higher (Cockgroft Gault formula).
* No concurrent illnesses that would prevent taking oral therapy and interfere with safety assessment.

Part 4 Eligibility Criterion:

- For subjects enrolling into Part 4 (PTCy/Tac/MMF), patients must have a left ventricular ejection fraction at least 45% within 3 months of first dose on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
MTD of Venetoclax with Busulfan and Fludarabine | 37 Days
  Determine safe dose and schedule of venetoclax
MTD of Venetoclax with Azacitidine as Maintenance Therapy | 28 Days from Maintenance Therapy Start
  Determine safe dose and schedule of venetoclax
MTD of Venetoclax with Decitabine/cedazuridine as Maintenance Therapy | 28 Days from Maintenance Therapy Start
  Determine safe dose and schedule of venetoclax

SECONDARY OUTCOMES:
Overall Survival | 12 Months
  Time from treatment start until death
Progression Free Survival | 12 Months
  Time from treatment start until relapse
Overall Response Rate | At day 100, 6 months and 12 months
  IWG response criteria
Remission Duration Rate | from start of the treatment until disease relapse (assessed at day 100, 6 months and 12 months)
  Duration of remission from treatment start until relapse
Rate of Disease Relapse | 12 Months
  Frequency of disease recurrence on trial
Rate of Non-Relapse Mortality | 12 Months
  Frequency of death that is not due to disease recurrence on trial
Donor granulocyte chimerism percentage | 28 Days Post-Transplant
  Percentage of donor blood cells
Donor granulocyte chimerism percentage | 100 days Post-Transplant
  Percentage of donor blood cells
Donor granulocyte chimerism percentage | 12 Months Post-Transplant
  Percentage of donor blood cells
Cumulative incidence of acute graft versus host disease (GVHD) and chronic GVHD following allo-HCT | 12 Months
  Frequency of GVHD events
Number of Maintenance Treatment Cycles Safely Administered | From Initiation of Maintenace Therapy up to 12 months
  Maintenance Treatment Cycles
Compare Incidences of Mortality and Survival Between Participants in Part 1, Part 2 and Part 3 | 12 months
  Compare cumulative instances of mortality and survival between participants on Part 1, Part 2 and Part 3

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline S. Garcia, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia JS, Kim HT, Murdock HM, Cutler CS, Brock J, Gooptu M, Ho VT, Koreth J, Nikiforow S, Romee R, Shapiro R, Loschi F, Ryan J, Fell G, Karp HQ, Lucas F, Kim AS, Potter D, Mashaka T, Stone RM, DeAngelo DJ, Letai A, Lindsley RC, Soiffer RJ, Antin JH. Adding venetoclax to fludarabine/busulfan RIC transplant for high-risk MDS and AML is feasible, safe, and active. Blood Adv. 2021 Dec 28;5(24):5536-5545. doi: 10.1182/bloodadvances.2021005566. PMID 34614506
- [Background] Garcia JS, Kim HT, Murdock HM, Ansuinelli M, Brock J, Cutler CS, Gooptu M, Ho VT, Koreth J, Nikiforow S, Romee R, Shapiro R, DeAngelo DJ, Stone RM, Bat-Erdene D, Ryan J, Contreras ME, Fell G, Letai A, Ritz J, Lindsley RC, Soiffer RJ, Antin JH. Prophylactic maintenance with venetoclax/azacitidine after reduced-intensity conditioning allogeneic transplant for high-risk MDS and AML. Blood Adv. 2024 Feb 27;8(4):978-990. doi: 10.1182/bloodadvances.2023012120. PMID 38197938
- [Derived] Garcia JS, Kim HT, Murdock HM, Bosch-Vilaseca A, Panaro KM, Lim F, Fiorilla J, Auriemma E, Brock J, Gooptu M, Ho VT, Cutler CS, Shapiro RM, Kelkar AH, Abel GA, DeAngelo DJ, Stone RM, Bat-Erdene D, Ryan JA, Fell G, Letai A, Ritz J, Lindsley RC, Antin JH, Soiffer RJ. Venetoclax/FluBu2 RIC transplant followed by all-oral venetoclax/decitabine maintenance for poor risk MDS/AML. Blood Adv. 2025 Dec 5:bloodadvances.2025018631. doi: 10.1182/bloodadvances.2025018631. Online ahead of print. PMID 41348911